CLINICAL TRIAL: NCT02514616
Title: Electrical Stimulation Therapy (EST) of the Lower Esophageal Sphincter: a Multicenter, Randomized, Double-blind, Sham-controlled Parallel-group Trial Evaluating Short Term Efficacy of EndoStim Device on GERD
Brief Title: Electrical Stimulation Therapy (EST) of the Lower Esophageal Sphincter (GERD)
Acronym: EST-SHAM-EUR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early termination due to a suspension of financial support
Sponsor: Erasme University Hospital (Other)
Collaborators: EndoStim Inc. (Industry)
Responsible Party: Principal Investigator, Hubert Louis, Hubert LOUIS, pHD, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ESE-001
Record Dates: First submitted 2015-07-24; First posted 2015-08-04 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: GERD
Keywords: Reflux; Reflux disease; Gastroesophageal reflux disease; Lower esophageal sphincter stimulation
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Electric Stimulation Therapy (Active Comparator): The subject receives Active Electric Stimulation Therapy for 12 weeks, 2 weeks after laparoscopic IPG and lead implant procedure. The subject and physician will be blinded to the randomization group assignment. The subject continues on stimulation treatment after 14 weeks and an extended open-label follow-up phase includes annual visits through 5 years.
  Interventions: Procedure: Laparoscopic IPG and lead implant procedure; Device: Active Electric Stimulation Therapy
- Delayed Electric Stimulation Therapy (Sham Comparator): The subject receives no active Electric Stimulation Therapy for 12 weeks, 2 weeks after laparoscopic IPG and lead implant procedure. The subject and physician will be blinded to the randomization group assignment. The subject will receive Active Electric Stimulation Therapy at week 14 visit, and an extended open-label follow-up phase includes annual visits through 5 years.
  Interventions: Procedure: Laparoscopic IPG and lead implant procedure; Device: Delayed Electric Stimulation Therapy

INTERVENTIONS:
Procedure: Laparoscopic IPG and lead implant procedure — EST placement
  Other Names: EndoStim
Device: Active Electric Stimulation Therapy — Device programming by the technician to deliver the EST system active (Treatment group) or no stimulation (Control group) for the following 12 weeks, at the 2 weeks visit.
  Other Names: EndoStim
  Arms: Active Electric Stimulation Therapy
Device: Delayed Electric Stimulation Therapy — Device programming by the technician to deliver the EST system no stimulation for the following 12 weeks at the 2 weeks visit. Active Electric Stimulation Therapy will be programmed at the 14 weeks visit.
  Other Names: EndoStim
  Arms: Delayed Electric Stimulation Therapy

SUMMARY:
The investigational device that will be used in this trial is the EndoStim® Lower Esophageal Sphincter (LES) Stimulation System.

The purpose of this trial is to evaluate the safety and the effectiveness of electrical stimulation therapy (EST) on the lower esophageal sphincter (LES) in the treatment of subjects with gastroesophageal reflux disease (GERD).

The study population will consist of subjects diagnosed with pathological GERD as defined by abnormal pH and who complain of heartburn, regurgitation or both for > 6 months, on a daily PPI use.

DETAILED DESCRIPTION:
Study Design:

Multicenter, randomized, double-blind, sham-controlled study. All subjects undergo screening and baseline visits, followed by system implantation, and randomization after 2 weeks to either a treatment Group (stimulation) or Control Group (delayed stimulation).

Randomized subjects complete a 10-week, double-blind phase. At the 14-week visit, subjects are unblinded, control group subjects begin receiving stimulation, and all subjects are followed for an additional 9-month open-label treatment phase.

Subjects continue receiving stimulation for an extended follow-up phase involving annual visits through 5 years.

Study Visits:

Screening and baseline visits. Laparoscopic implantable pulse generator (IPG) and lead implant procedure. Post-implant follow-up office visits at 2 weeks/randomization, 6, 10, 14, 24 and 48 weeks, followed by annual visits through 5 years.

Sample Size and Scope:

Forty-six subjects will be implanted and followed to 12 months after stimulation treatment at 3 investigational sites.

ELIGIBILITY:
Inclusion Criteria:

* Subject able and willing to provide written informed consent
* Subject able and willing to comply with required study procedures and follow-up schedule
* Typical symptoms of GERD (regurgitation and/or heartburn) for longer than 6 months, heartburn responding to PPI therapy. Subject may also complain of atypical symptoms of GERD that may persist on PPI
* Daily dose of PPI or other acid neutralization drugs because of PPI intolerance
* Baseline visit GERD-HRQL score ≥ 20 following 14 days off-PPI and at least 10 points higher than their on-PPI (or other acid-neutralization drugs) GERD-HRQL score recorded during the Screening Visit
* Excessive lower esophageal acid exposure during pH monitoring (defined as distal esophageal pH < 4 for > 5.0% of the monitoring time) performed after 14 days off PPIs
* Subject is a suitable surgical candidate able to undergo general anesthesia and laparoscopic surgery.

Exclusion Criteria:

* Previous EndoStim LES System implant and/or implant attempt
* Previous esophageal surgery, including Nissen fundoplication
* Previous endoscopic intervention for the treatment of GERD and/or Barrett's esophagus
* Hiatal hernia larger than 2 cm as determined by any diagnostic investigation (i.e., endoscopy, manometry or laparoscopic visualization)
* Gastroparesis
* Any non-GERD esophageal motility disorders
* Esophageal stricture or significant esophageal anatomic abnormalities
* Barrett's epithelium or any grade of dysplasia
* Documented history of esophagitis Grade C or D (LA Classification)
* History of suspected or confirmed esophageal or gastric cancer
* Esophageal or gastric varices
* Symptoms of dysphagia more than once per week within the last 3 months
* Suspected or known allergies to titanium, platinum, iridium, stainless steel, silicone, epoxy, or nylon
* Body mass index (BMI) > 35 kg/m2
* Any significant multisystem diseases
* Autoimmune or a connective tissue disorder (scleroderma, dermatomyositis, Calcinosis-Raynaud's-Esophagus Sclerodactyly Syndrome (CREST), Sjogren's Syndrome, Sharp's Syndrome, etc.) requiring therapy in the preceding 2 years
* Type 1 diabetes mellitus or uncontrolled Type 2 diabetes mellitus (T2DM) defined as HbA1c > 9.5 in the previous 6 months or at screening/baseline, or has T2DM for > 10 years
* Significant cardiac arrhythmia or ectopy or significant cardiovascular disease (i.e. unstable angina pectoris, hemodynamically significant valvular disease, severe congestive heart failure), or cardiac therapeutic intervention within the last 6 months.
* Significant cerebrovascular event within the last 6 months
* Existing implanted electrical stimulator (pacemaker, implantable cardioverter defibrillator, deep brain stimulator (DBS), bone growth or pelvic floor stimulators, drug pumps, etc.)
* Chronic anticoagulant therapy
* Female subject of child-bearing potential and is pregnant or nursing, or intends to become pregnant during the trial period, who is not using a reliable form of birth control
* Subject is currently enrolled in other potentially confounding research
* Active infection as determined by the investigator
* History of any malignancy in the last 2 years
* Life expectancy less than 3 years
* Diagnosed major psychiatric disorder (bipolar, schizophrenia, etc.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of EST on GERD symptoms (mean improvement in the GERD- health-related quality of life (HRQL) scores from baseline in control and treatment groups) | 14 weeks
  Comparison between Treatment and Control Groups of the mean improvement in the composite GERD-HRQL scores from baseline measured after at least 14 days off proton pump inhibitors (PPIs)

SECONDARY OUTCOMES:
Safety (Rate of occurrence of device- and procedure-related adverse events) | 12 months
Number of subjects achieving GERD symptom success | 12 months
  Improvement in the total GERD-HRQL score of 50% or more compared to pre-implantation score off PPI
Reflux symptoms measured by GERD-HRQL score | 6 months
  Mean improvement in the composite GERD-HRQL scores from baseline measured after at least 14 days off proton pump inhibitors (PPIs)
Reflux symptoms measured by GERD-HRQL score | 12 months
  Mean improvement in the composite GERD-HRQL scores from baseline measured after at least 14 days off proton pump inhibitors (PPIs)
Number of subjects able to stop regular use of acid-suppression | 12 months
  Defined as 50% or more days without PPI use
Number of subjects able to stop all use of acid-suppression medication | 12 months
Percentage of asymptomatic patients | 14 weeks
  Defined as an improvement in their total GERD-HRQL score of 50% or more compared to pre-implantation score off PPI) in treatment and control groups, off-PPI for the last 2 weeks.
Incidence of reflux esophagitis | 12 months
Quality of life measured by EQ-5D EuroQol score | 14 weeks
  Difference in patient's EQ-5D score, compared to pre-implantation score on and off PPI.
Quality of life measured by EQ-5D score | 6 months
  Difference in patient's EQ-5D score, compared to pre-implantation score on and off PPI.
Quality of life measured by EQ-5D score | 12 months
  Difference in patient's EQ-5D score, compared to pre-implantation score on and off PPI.
Efficacy of EST on acid reflux measured by esophageal pH | 14 weeks
  Difference in % 24 hour esophageal pH<4 in Treatment and Control groups (total, upright, supine, postprandial (2h)).
Efficacy of EST on acid reflux measured by DeMeester score | 14 weeks
  Difference in DeMeester score in Treatment and Control groups.
Percentage of subjects achieving pH success | 14 weeks
  Defined as normalization (pH < 4 for no more than 4.1% of monitoring time) or > 50% improvement in their distal esophageal acid exposure compared to their baseline off-PPI distal esophageal pH.
Efficacy of EST on reflux episodes measured by esophageal impedance | 14 weeks
  Difference in the number of reflux episodes (total, upright, supine, postprandial (2h), acidic, weakly acidic, weakly alkaline, and proximal extent (15 cm) in Treatment and Control groups.
Difference in lower esophageal sphincter (LOS) pressure and integrated relaxation pressure at 4 seconds (IRP4s) in Treatment and Control groups | 14 weeks
Comparison of GERD-HRQL scores in Treatment and Control groups | 14 weeks
Comparison of quality of life measured by EQ-5D in Treatment and Control groups | 14 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Gastroenterology Department, Erasme University Hospital, Brussels, Belgium
- Hôpital Edouard Herriot, Service d'Explorations Fonctionnelles Digestives, Pavillons H et L, 5 Place d'Arsonval, Lyon, Lyon Cedex 3, France